CLINICAL TRIAL: NCT04610996
Title: The Validation of Calculated Equations of GFR in Thai Chronic Kidney Disease
Brief Title: The Valid of GFR in Chronic Kidney Disease Patients
Status: Withdrawn | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Other Study IDs: RVH-CR-002; Rajavithi Hospital
Record Dates: First submitted 2008-08-02; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Chronic Kidney Disease
Keywords: GFR CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study was cancel due to principle investigator had been resigned

DETAILED DESCRIPTION:
Study was cancel due to principle investigator had been resigned

ELIGIBILITY:
Inclusion Criteria:

* Age more than 16

Exclusion Criteria:

* none

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population in Dindang Destric, central Bangkok regoin was select in this cohort.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-09 (Actual)